CLINICAL TRIAL: NCT00806962
Title: Randomized Double-Blind Placebo-Controlled Phase 1, Safety and Immunogenicity Study of Two Dosages of Intranasal Norwalk Virus-like Particle Vaccine ( Norwalk VLP Antigen, MPL®, Chitosan, Mannitol, and Sucrose) Compared to Adjuvant/Excipients (MPL®, Chitosan, Mannitol, and Sucrose) and to Placebo (Empty Device
Brief Title: Phase 1 Norwalk Vaccine Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LigoCyte Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LV01-102
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Norovirus
MeSH Terms: interventions — Adjuvants, Pharmaceutic; Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vaccine Arm 1 (Experimental): 50 µg Norwalk VLP Vaccine + Adjuvant/Excipients
  Interventions: Biological: Norwalk VLP Vaccine
- Vaccine Arm 2 (Experimental): 100 µg Norwalk VLP Vaccine + Adjuvant/Excipients
  Interventions: Biological: Norwalk VLP Vaccine
- Adjuvant/Excipients (MPL) (Active Comparator): 14 mg chitosan, 3 mg mannitol, 3 mg sucrose, and 50 mcg MPL
  Interventions: Drug: Adjuvant/Excipients
- Empty device (Sham Comparator): Empty device that contains no dry powder formulation. Actuation of the empty intranasal delivery device will deliver a puff of air per device.
  Interventions: Device: placebo

INTERVENTIONS:
Drug: Adjuvant/Excipients — intranasal,14 mg chitosan, 3 mg mannitol, 3 mg sucrose and 50 mcg of MPL, 2 doses 21 days apart
  Arms: Adjuvant/Excipients (MPL)
Device: placebo — intranasal, puff of air, 2 doses, 21 days apart
  Arms: Empty device
Biological: Norwalk VLP Vaccine — intranasal, 50mcg, 2 doses--21 days apart
  Arms: Vaccine Arm 1
Biological: Norwalk VLP Vaccine — Intranasal, 100 mcg, 2 doses, 21 days apart
  Arms: Vaccine Arm 2

SUMMARY:
Randomized, double blind, multi-site, study in healthy adults, comparing safety and immunogenicity of two dosage levels of Norwalk VLP Vaccine with adjuvant/excipients and with placebo controls

Primary Objective:

* Safety as determined by occurrence of local intranasal symptoms or other symptoms as reported by a self-administered memory aid for 7 days after each vaccination and hematology, blood chemistry and physical examinations performed by the clinical research staff
* Subjects will also be monitored for Serious Adverse Events (SAEs), and onset of any new medical conditions for 180 days following the last study vaccinations (Day 201).

Secondary Objectives

Evaluations of immunogenicity as determined by:

* Geometric mean titers and seroconversion rate of serum anti- Norwalk VLP IgG and IgA
* Stimulation of anti-Norwalk VLP IgA antibody secreting cells (ASC)
* Presence of antigen specific memory B-cell response

Cells will be collected and stored for possible future evaluation of Norwalk VLP-specific cell-mediated immune (CMI) responses

Study Hypothesis:

The incidence of adverse events after intranasal Norwalk VLP Vaccine will be the same as the incidence of adverse events after intranasal adjuvant/excipients alone. Norwalk VLP Vaccine and adjuvant/excipients will have a higher incidence of mild to moderate nasal adverse events compared to placebo but similar incidence of other adverse events.

Two doses of the 100 µg of Norwalk VLP Vaccine will be more immunogenic than two doses of 50 µg of Norwalk VLP Vaccine. The post-vaccination serum antibody responses, the number of antibody secreting cells (ASC) and IgG and IgA memory B-cell responses directed against Norwalk Virus antigen will be increased after Norwalk VLP Vaccine compared to adjuvant/excipients and to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age 18 - 50 years, inclusive
3. Good general health as determined by a screening evaluation within 30 days before administration of Norwalk VLP Vaccine, adjuvant/excipients or placebo
4. Expressed interest and availability to fulfill the study requirements
5. Agrees not to become pregnant from the time of study enrollment until at least 56 days after the last administration of Norwalk VLP Vaccine, adjuvant/excipients or placebo; if a woman is sexually active and capable of conception (i.e., no history of hysterectomy or tubal ligation), she must agree to use hormonal or barrier birth control. A woman is eligible if she is monogamous with a male who has had a vasectomy.
6. Demonstrated to be an H type-1 antigen secretor
7. Agrees not to participate in another clinical trial with an investigational product for the entire duration of the study (six months after the last study dose i.e. 201 days)
8. Agrees to storage of unused clinical specimens for an indefinite period of time only for those specimens collected by the University of Maryland CVD for use in future research at the CVD. [A University of Maryland site-specific inclusion criterion]

Exclusion Criteria

1. History of any of the following medical illnesses

   * Chronic rhinitis, runny nose, sneezing
   * Clinically significant nose bleed within the last year
   * Diabetes
   * Cancer
   * Heart disease (hospitalization for a heart attack, arrhythmia, or syncope)
   * Unconsciousness (other than a single brief "concussion")
   * Seizures (other than febrile seizures as a child <5 years old)
   * Recurrent infections (more than 3 hospitalizations for invasive bacterial infections such as pneumonia or meningitis)
   * Asthma requiring treatment with inhaler or medication
   * Any current illness requiring daily medication other than vitamins, birth control, or anti-depressant
2. Blood Type B or AB, regardless of Rh + or -
3. Allergies or hypersensitivity to chitosan, shrimp, other shellfish or any component of the vaccine, adjuvant/excipients or placebo
4. History of nasal surgery of any type (including tonsilectomy/adenoidectomy)
5. Any clinically significant abnormality detected on physical examination, including:

   * Murmur (other than a functional murmur)
   * Focal neurological abnormality
   * Hepatosplenomegaly
   * Lymphadenopathy
   * Jaundice
6. Hypertension (BP > 140/90 mm Hg on two separate days)
7. Any lab abnormality, as listed below:

   * Neutrophils (WBC) outside the normal range
   * Hemoglobin outside the normal range (may be repeated once if outside this limit)
   * Platelet count outside the normal range (may be repeated once if outside this limit)
   * Creatinine outside the normal range (may be repeated once if outside this limit)
   * Glucose > upper limit of normal (may be repeated once if outside this limit)
   * AST or ALT outside the normal range (may be repeated once if outside this limit)
   * Positive serology for hepatitis C or HIV antibody or hepatitis B surface antigen
8. For women, positive serum pregnancy test within 7 days and urine pregnancy test within 24 hours of administering either dose of Norwalk VLP Vaccine, adjuvant/excipients or placebo
9. Nursing mother
10. Temperature > 38.0 degrees C (100.4 degrees F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 3 days of administration of Norwalk VLP Vaccine, adjuvant/excipients or placebo
11. Previous participation in a study of Norovirus vaccines
12. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
13. Receipt of an investigational vaccine or drug within 28 days before administration of Norwalk VLP Vaccine, adjuvant/excipients or placebo
14. Other condition that in the clinical judgment of the investigator would jeopardize the safety or rights of a subject participating in the trial, would render the subject unable to comply with the protocol or would interfere with the evaluation of the vaccine
15. Failure to pass written examination about this study (70% correct answers required to pass)[A University of Maryland site-specific exclusion criterion]

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
adverse events | seven days

SECONDARY OUTCOMES:
immunogenicity | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John J Treanor, MD, Principal Investigator — University of Rochester
Locations (4):
- United States (4):
  - University of Maryland Center for Vaccine Development, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio

REFERENCES:
- [Derived] El-Kamary SS, Pasetti MF, Mendelman PM, Frey SE, Bernstein DI, Treanor JJ, Ferreira J, Chen WH, Sublett R, Richardson C, Bargatze RF, Sztein MB, Tacket CO. Adjuvanted intranasal Norwalk virus-like particle vaccine elicits antibodies and antibody-secreting cells that express homing receptors for mucosal and peripheral lymphoid tissues. J Infect Dis. 2010 Dec 1;202(11):1649-58. doi: 10.1086/657087. Epub 2010 Oct 27. PMID 20979455